CLINICAL TRIAL: NCT00591006
Title: Phenytoin as a Neuroprotective Agent Against Corticosteroid-induced Functional Imaging Changes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Sherwood Brown, Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1R21MH078182 (NIH)
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Results first posted 2015-08-19 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: Phenytoin; Dilantin; Corticosteroid; Neuroprotection; Mania; Cognition; Mood; Memory; Hydrocortisone; Healthy Controls; MRI; hippocampal activation
MeSH Terms: conditions — Mania | interventions — Phenytoin; Hydrocortisone; Adrenal Cortex Hormones; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Four Treatments Per Participant (Experimental): This study has one arm due to a crossover design. All 17 subjects received 4 treatments: placebo then placebo, phenytoin then placebo, placebo then hydrocortisone, and phenytoin then hydrocortisone. Each treatment was randomly assigned and had a unique sequence out of 24 possible sequences.
  Interventions: Drug: Phenytoin (brand name Dilantin); Drug: Hydrocortisone; Drug: Placebo

INTERVENTIONS:
Drug: Phenytoin (brand name Dilantin) — Three days prior to imaging, participants will take two capsules containing phenytoin tablets (100 mg) by mouth at 0900 hours and 2100 hours (400 mg/day) for a total of three days with the last dose at 0900 hours on the day of the imaging (7 doses total).
  Other Names: 5,5-Diphenylhydantoin; Fenitoin; Antisacer; Difenin; Dihydan; Dilantin; Diphenylhydantoin; Epamin; Hydantol; Sodium Diphenylhydantoinate
Drug: Hydrocortisone — Beginning two days prior to the imaging (the day after initiating the phenytoin or placebo), participants will begin taking 4 tablets containing hydrocortisone (20 mg) or placebo also at 0900 hours and 2100 hours (160 mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The doses were selected to achieve a low therapeutic blood level of phenytoin and stress level of cortisol. Newcomer et al. (1999) used this dose of hydrocortisone in healthy controls. The imaging will be performed at approximately 1300 hours.
  Other Names: Cortef; Corticosteroids
Drug: Placebo — Participants take two capsules of placebo 100 mg at 0900 hours and 2100 hours for a total of 3 days with the last dose at 0900 hours on the day of imaging (7 doses total). Beginning two days prior to the imaging (the day after initiating placebo), participants will being taking 4 tablets containing placebo (20 mg) also at 0900 hours and 2100 hours with the last dose at 0900 hours on the day of the imaging (5 doses total).
  Other Names: Sugar pill

SUMMARY:
The purpose of this research is to determine if patients who receive phenytoin (also commonly known as Dilantin) before taking corticosteroids will show less memory impairment and hypomanic symptoms (feelings of agitation, overexcitement or hyperactivity) than those receiving placebo (an inactive substance). This research also seeks to determine if patients taking phenytoin before corticosteroids show more activity in the area of the brain involved with memory than those receiving placebo.

This research is being done because increased levels of cortisol (the body's natural corticosteroid) in the body are frequently associated with forgetfulness, and interventions that may prevent or reverse this effect are of great importance.

DETAILED DESCRIPTION:
Introduction and aims: Stress and corticosteroid exposure are associated with changes in the human and animal hippocampus. In animals, phenytoin prevents dendritic changes in the hippocampus secondary to corticosterone. We propose to use functional magnetic resonance imaging (fMRI) to explore the effects of 3-days of exposure to placebo, hydrocortisone, phenytoin and hydrocortisone plus phenytoin on hippocampal activation. If phenytoin attenuates the effects of hydrocortisone, we will use this model system to explore other potential neuroprotective agents

CONCISE SUMMARY OF PROJECT: Sixteen healthy participants will, in a one-hour imaging session, receive a structural magnetic resonance imaging (MRI), magnetic resonance spectroscopy (MRS) and fMRI scan four separate times with a 21 day washout between each study drug exposure in a crossover design. Prior to each scan each participant will receive placebo + placebo, phenytoin + placebo, hydrocortisone + placebo, or hydrocortisone + phenytoin in a random fashion. Thus, each participant will receive each of the four possible study drug combinations in a random order with an extended drug washout between each exposure. Hippocampal activation, volume and biochemistry, as well as mood and memory will be assessed. The figure in Appendix I illustrates the study design.

All participants will complete a University of Texas (UT) Southwestern (UTSW) Institutional Review Board (IRB) approved informed consent process and give written consent to participate prior to study entry.

At the first screening visit, demographic information and a complete medical and psychiatric history will be obtained. The Structured Clinical Interview for DSM-IV (SCID) (First et al 1995) will be used to rule out exclusionary psychiatric illnesses. Mood will be assessed with the Hamilton Rating Scale for Depression (HRSD), Young Mania Rating Scale (YMRS), and Activation (ACT) subscale of the ISS. Cognition will be assessed with the Rey Auditory Verbal Learning Test (RAVLT) (declarative memory-hippocampus), Digit Span Backwards, and two computer tests - the Sternberg Memory Task (SMT, declarative memory-hippocampus) (Sternberg 1969), and Running Memory Continuous Performance Task (RMCPT, working memory-prefrontal cortex) (Baddeley 1986). Alternative versions of the tests will be used throughout the study to minimize any learning effects. For subjects who successfully pass the screening, fMRI sessions will be scheduled, and they will be asked to return 4 days prior to their first scan. If subjects feel uncomfortable answering any questions on the questionnaires during their screening visit, they can refuse to do so, and they will be removed from the study. If any psychological disorders are diagnosed at this stage (e.g., mood disorders such as depression), subjects will be removed from the study and referred either to Parkland hospital or to a private psychiatrist based on their insurance coverage for further evaluations and treatment. If at a later stage any abnormalities are uncovered through imaging, subjects will be notified immediately. Subjects will be provided with a referral to either Parkland Hospital or a different facility based on their insurance coverage. With the subject's consent, we will also notify their primary physician. Pregnancy tests will be obtained for females at baseline and prior to the start of each new medication cycle to ensure that no pregnant women are participating in the study (5 times total during the study).

One day prior to each study drug course, mood will be assessed with HRSD, YMRS, and ACT subscale of Internal State Scale, and cognition will be assessed with the Sternberg Memory Task.

Three days prior to imaging, participants will take two capsules containing phenytoin tablets (100 mg) or identical placebo by mouth at 0900 hours and 2100 hours (400 mg/day) for a total of three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Beginning two days prior to the imaging (the day after initiating the phenytoin or placebo), participants will begin taking 4 tablets containing hydrocortisone (20 mg) or placebo also at 0900 hours and 2100 hours (160 mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The doses were selected to achieve a low therapeutic blood level of phenytoin and stress level of cortisol. Newcomer et al. (1999) used this dose of hydrocortisone in healthy controls. The imaging will be performed at approximately 1300 hours.

Imaging will be performed after each three day exposure to study medications. Mood assessments and the SMT will be conducted at baseline and prior to and after each course of study medication (day medication course begins and on the day of the neuroimaging). The SMT has a large number of equivalent versions and thus can be administered numerous times. By administering prior to each exposure to study drug we can determine whether or not memory will, as expected, have returned to baseline after each washout period. Other cognitive testing including the RAVLT, Digits Backwards, and RMCPT will be performed after each course of study medication. Cognitive testing is not performed prior to receiving the study medication to avoid multiple testing over a short period of time which is unnecessary given the baseline and placebo data which can be used for comparison.

Monitoring study drug levels: Blood will be drawn at baseline (approximately 1400 hours) to assess cortisol levels. Blood will be drawn after each scan (approximately 1400 hours) to assess cortisol and phenytoin levels and to ensure adherence to the medications. We anticipate an increase in cortisol levels following administration of cortisol compared to baseline in subjects taking cortisol, and that therapeutic levels of phenytoin for seizures (10 to 20 mg/l) will be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Men or women
* Vision corrected to at least 20-40
* No tobacco use
* Education of ≥12 years (No GED)

Exclusion Criteria:

* History of major psychiatric illness defined as major depressive disorder, bipolar disorder, post traumatic stress disorder, panic disorder, schizoaffective disorder, schizophrenia or eating disorders
* History of drug or alcohol abuse or dependence
* History of neurological disorders including seizures, brain surgery, multiple sclerosis, Parkinson's disease
* Taking central nervous system (CNS) acting medications (e.g. antidepressants, hypnotics)
* History of allergic reaction or medical contraindication to phenytoin or hydrocortisone therapy
* Metal implants, claustrophobia or other contraindications to MRI
* Significant medical conditions (e.g. myocardial infarction, diabetes)
* Pregnant or nursing women
* Prisoners
* History of mental retardation, special education classes, dementia or other severe cognitive disorders
* Baseline Hamilton Rating Scale for Depression Score > 7
* History of a suicide attempt
* History of systemic corticosteroid use or current inhaled corticosteroid use

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2008-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherwood Brown, M.D.,Ph.D., Principal Investigator — UT Southwestern Medical Center of Dallas
Locations (1):
- UT Southwestern Medical Center of Dallas/Parkland Memorial Hospital, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began 3/11/2008 and was completed 4/23/2009. Subjects were recruited through flyers posted at UTSW medical clinics.
Pre-assignment Details: Subjects were enrolled and randomized to one out of 4 treatments. The study design is a 4-phase crossover study, meaning all subjects received all four treatments during the course of the study. Subjects washed out of each medication cycle for 21 days before beginning the next treatment cycle. Total number of subjects enrolled is 17.
Groups:
- PH + PL Then PL + H Then PL + H Then PL + PL: Participants take two capsules containing phenytoin tablets by mouth at 0900 hours and 2100 hours (400 mg/day) for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the phenytoin), participants will begin taking 4 tablets containing placebo also at 0900 hours and 2100 hours with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking phenytoin tablets followed by hydrocortisone (160 mg/day). The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take placebo followed by hydrocortisone. The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take placebo followed by placebo. The imaging will be performed at 1300 hours.
- PH + H Then PH + PL Then PL + H Then PL + PL: Participants take two capsules containing phenytoin tablets by mouth at 0900 hours and 2100 hours (400 mg/day) for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the phenytoin), participants will begin taking 4 tablets containing hydrocortisone also at 0900 hours and 2100 hours (160 mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking phenytoin tablets followed by placebo. The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take placebo followed by hydrocortisone. The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take placebo followed by placebo. The imaging will be performed at 1300 hours.
- PL + PL Then PH + PL Then PH + H Then PL + H: Participants take two capsules containing placebo tablets by mouth at 0900 hours and 2100 hours for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the placebo), participants will begin taking 4 tablets containing placebo also at 0900 hours and 2100 hours with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking phenytoin tablets (400mg/day) followed by placebo. The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take phenytoin followed by hydrocortisone (160mg/day). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take placebo followed by hydrocortisone. The imaging will be performed at 1300 hours.
- PL + H Then PL + PL Then PH + PL Then PH + H: Participants take two capsules containing placebo tablets by mouth at 0900 hours and 2100 hours for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the placebo), participants will begin taking 4 tablets containing hydrocortisone also at 0900 hours (20mg) and 2100 hours (160mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking placebo tablets followed by placebo. The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take phenytoin (400mg/day) followed by hydrocortisone. The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take phenytoin followed by hydrocortisone. The imaging will be performed at 1300 hours.
- PL + H Then PH + PL Then PL + PL Then PH + H: Participants take two capsules containing placebo tablets by mouth at 0900 hours and 2100 hours for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the placebo), participants will begin taking 4 tablets containing hydrocortisone also at 0900 hours and 2100 hours (160mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking phenytoin tablets (400mg/day) followed by placebo. The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take placebo followed by placebo. The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take phenytoin followed by hydrocortisone. The imaging will be performed at 1300 hours.
- PL + H Then PL + PL Then PH + H Then PH + PL: Participants take two capsules containing placebo tablets by mouth at 0900 hours and 2100 hours for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the placebo), participants will begin taking 4 tablets containing hydrocortisone also at 0900 hours and 2100 hours (160mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking placebo tablets followed by placebo. The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take phenytoin (400mg/day) followed by hydrocortisone. The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take phenytoin followed by placebo. The imaging will be performed at 1300 hours.
- PL + H Then PH +H Then PH + PL Then PL + PL: Participants take two capsules containing placebo tablets by mouth at 0900 hours and 2100 hours for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the placebo), participants will begin taking 4 tablets containing hydrocortisone also at 0900 hours and 2100 hours (160mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking phenytoin tablets (400mg/day) followed by hydrocortisone. The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take phenytoin followed by placebo. The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take placebo followed by placebo. The imaging will be performed at 1300 hours.
- PL + H Then PH + H Then PL + PL Then PH + PL: Participants take two capsules containing placebo tablets by mouth at 0900 hours and 2100 hours for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the placebo), participants will begin taking 4 tablets containing hydrocortisone also at 0900 hours and 2100 hours (160mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking phenytoin tablets (400mg/day) followed by hydrocortisone. The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take placebo followed by placebo. The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take phenytoin followed by placebo. The imaging will be performed at 1300 hours.
- PL + H Then PH + PL Then PH + H Then PL + PL: Participants take two capsules containing placebo tablets by mouth at 0900 hours and 2100 hours for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the placebo), participants will begin taking 4 tablets containing hydrocortisone also at 0900 hours and 2100 hours (160mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking phenytoin tablets (400mg/day) followed by placebo. The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take phenytoin followed by hydrocortisone. The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take placebo followed by placebo. The imaging will be performed at 1300 hours.
- PH + H Then PL + H Then PL + PL Then PH + PL: Participants take two capsules containing phenytoin tablets by mouth at 0900 hours and 2100 hours (400mg/day) for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the phenytoin), participants will begin taking 4 tablets containing hydrocortisone also at 0900 hours and 2100 hours (160mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking placebo tablets followed by hydrocortisone. The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take placebo followed by placebo. The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take phenytoin followed by placebo. The imaging will be performed at 1300 hours.
- PH + H Then PL + H Then PH + PL Then PL + PL: Participants take two capsules containing phenytoin tablets by mouth at 0900 hours and 2100 hours (400mg/day) for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the phenytoin), participants will begin taking 4 tablets containing hydrocortisone also at 0900 hours and 2100 hours (160mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking placebo tablets followed by hydrocortisone. The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take phenytoin followed by placebo. The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take placebo followed by placebo. The imaging will be performed at 1300 hours.
- PH + H Then PH + PL Then PL + PL Then PL + H: Participants take two capsules containing phenytoin tablets by mouth at 0900 hours and 2100 hours (400mg/day) for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the phenytoin), participants will begin taking 4 tablets containing hydrocortisone also at 0900 hours and 2100 hours (160mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking phenytoin tablets followed by placebo. The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take placebo followed by placebo. The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take placebo followed by hydrocortisone. The imaging will be performed at 1300 hours.
- PH + H Then PL + PL Then PH + PL Then PL + H: Participants take two capsules containing phenytoin tablets by mouth at 0900 hours and 2100 hours (400mg/day) for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the phenytoin), participants will begin taking 4 tablets containing hydrocortisone also at 0900 hours and 2100 hours (160mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking placebo tablets followed by placebo. The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take phenytoin followed by placebo. The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take placebo followed by hydrocortisone. The imaging will be performed at 1300 hours.
- PH + H Then PL + PL Then PL + H Then PH + PL: Participants take two capsules containing phenytoin tablets by mouth at 0900 hours and 2100 hours (400mg/day) for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the phenytoin), participants will begin taking 4 tablets containing hydrocortisone also at 0900 hours and 2100 hours (160mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking placebo tablets followed by placebo. The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take placebo followed by hydrocortisone. The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take phenytoin followed by placebo. The imaging will be performed at 1300 hours.
- PH + PL Then PL + PL Then PH + H Then PL + H: Participants take two capsules containing phenytoin tablets by mouth at 0900 hours and 2100 hours (400mg/day) for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the phenytoin), participants will begin taking 4 tablets containing placebo also at 0900 hours and 2100 hours with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking placebo tablets followed by placebo. The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take phenytoin followed by hydrocortisone (160mg/day). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take placebo followed by hydrocortisone. The imaging will be performed at 1300 hours.
- PH + PL Then PL + PL Then PL + H Then PH + H: Participants take two capsules containing phenytoin tablets by mouth at 0900 hours and 2100 hours (400mg/day) for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the phenytoin), participants will begin taking 4 tablets containing placebo also at 0900 hours and 2100 hours with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking placebo tablets followed by placebo. The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take placebo followed by hydrocortisone (160mg/day). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take phenytoin followed by hydrocortisone. The imaging will be performed at 1300 hours.
- PH + PL Then PH + H Then PL + PL Then PL + H: Participants take two capsules containing phenytoin tablets by mouth at 0900 hours and 2100 hours (400mg/day) for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the phenytoin), participants will begin taking 4 tablets containing placebo also at 0900 hours and 2100 hours with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking phenytoin tablets followed by hydrocortisone (160mg/day). The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take placebo followed by placebo. The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take placebo followed by hydrocortisone. The imaging will be performed at 1300 hours.
- PH + PL Then PH + H Then PL + H Then PL + PL: Participants take two capsules containing phenytoin tablets by mouth at 0900 hours and 2100 hours (400mg/day) for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the phenytoin), participants will begin taking 4 tablets containing placebo also at 0900 hours and 2100 hours with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking phenytoin followed by hydrocortisone (160mg/day). The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take placebo followed by hydrocortisone. The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take placebo followed by placebo. The imaging will be performed at 1300 hours.
- PL + PL Then PH + PL Then PL + H Then PH + H: Participants take two capsules containing placebo tablets by mouth at 0900 hours and 2100 hours for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the placebo), participants will begin taking 4 tablets containing placebo also at 0900 hours and 2100 hours with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking phenytoin tablets (400mg/day) followed by placebo. The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take placebo followed by hydrocortisone (160mg/day). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take phenytoin followed by hydrocortisone. The imaging will be performed at 1300 hours.
- PL + PL Then PH + H Then PH + PL Then PL + H: Participants take two capsules containing placebo tablets by mouth at 0900 hours and 2100 hours for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the placebo), participants will begin taking 4 tablets containing placebo also at 0900 hours and 2100 hours with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking phenytoin tablets (400mg/day) followed by hydrocortisone (160mg/day). The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take phenytoin followed by placebo. The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take placebo followed by hydrocortisone. The imaging will be performed at 1300 hours.
- PL + PL Then PL + H Then PH + PL Then PH + H: Participants take two capsules containing placebo tablets by mouth at 0900 hours and 2100 hours for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the placebo), participants will begin taking 4 tablets containing placebo also at 0900 hours and 2100 hours with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking placebo tablets followed by hydrocortisone (160mg/day). The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take phenytoin (400mg/day) followed by placebo. The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take phenytoin followed by hydrocortisone. The imaging will be performed at 1300 hours.
- PL + PL Then PL + H Then PH + H Then PH + PL: Participants take two capsules containing placebo tablets by mouth at 0900 hours and 2100 hours for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the placebo), participants will begin taking 4 tablets containing placebo also at 0900 hours and 2100 hours with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking placebo tablets followed by hydrocortisone (160mg/day). The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take phenytoin (400mg/day) followed by hydrocortisone. The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take phenytoin followed by placebo. The imaging will be performed at 1300 hours.
- PL + PL Then PH + H Then PL + H Then PH + PL: Participants take two capsules containing placebo tablets by mouth at 0900 hours and 2100 hours for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the placebo), participants will begin taking 4 tablets containing placebo also at 0900 hours and 2100 hours with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking phenytoin tablets (400mg/day) followed by hydrocortisone (160mg/day). The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take placebo followed by hydrocortisone. The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take phenytoin followed by placebo. The imaging will be performed at 1300 hours.
- PH + PL Then PL + H Then PL + PL Then PH + H: Participants take two capsules containing phenytoin tablets by mouth at 0900 hours and 2100 hours (400 mg/day) for three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Two days prior to the imaging (the day after initiating the phenytoin), participants will begin taking 4 tablets containing placebo also at 0900 hours and 2100 hours with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will repeat this cycle, instead taking placebo tablets followed by hydrocortisone (160mg/day). The imaging will be performed at 1300 hours and participants washout for 21 days. Participants then take placebo followed by placebo. The imaging will be performed at 1300 hours. Participants washout for 21 days. Participants will then take phenytoin followed by hydrocortisone. The imaging will be performed at 1300 hours.
Period: Overall Study
Arm/Group | PH + PL Then PL + H Then PL + H Then PL + PL | PH + H Then PH + PL Then PL + H Then PL + PL | PL + PL Then PH + PL Then PH + H Then PL + H | PL + H Then PL + PL Then PH + PL Then PH + H | PL + H Then PH + PL Then PL + PL Then PH + H | PL + H Then PL + PL Then PH + H Then PH + PL | PL + H Then PH +H Then PH + PL Then PL + PL | PL + H Then PH + H Then PL + PL Then PH + PL | PL + H Then PH + PL Then PH + H Then PL + PL | PH + H Then PL + H Then PL + PL Then PH + PL | PH + H Then PL + H Then PH + PL Then PL + PL | PH + H Then PH + PL Then PL + PL Then PL + H | PH + H Then PL + PL Then PH + PL Then PL + H | PH + H Then PL + PL Then PL + H Then PH + PL | PH + PL Then PL + PL Then PH + H Then PL + H | PH + PL Then PL + PL Then PL + H Then PH + H | PH + PL Then PH + H Then PL + PL Then PL + H | PH + PL Then PH + H Then PL + H Then PL + PL | PL + PL Then PH + PL Then PL + H Then PH + H | PL + PL Then PH + H Then PH + PL Then PL + H | PL + PL Then PL + H Then PH + PL Then PH + H | PL + PL Then PL + H Then PH + H Then PH + PL | PL + PL Then PH + H Then PL + H Then PH + PL | PH + PL Then PL + H Then PL + PL Then PH + H
Started | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1
Treatment #2 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1
Treatment #3 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1
Treatment #4 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Completed | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Study Population: Seventeen healthy controls, in a one-hour imaging session, received a structural MRI, MRS and fMRI scan four separate times with a 21 day washout between each study drug exposure in a crossover design. Prior to each scan each participant received placebo + placebo, phenytoin + placebo, hydrocortisone + placebo, or hydrocortisone + phenytoin in a random fashion. Thus, each participant received each of the four possible study drug combinations in a random order with an extended drug washout between each exposure. Hippocampal activation, volume and biochemistry, as well as mood and memory was assessed.
Arm/Group | Total Study Population
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Difference in RAVLT Total T-Score Between Treatments
Description: The Rey Auditory Verbal Learning Test (RAVLT) evaluates a wide diversity of functions, including short-term auditory-verbal memory, and retention of information. Test raw scores are converted to T-scores. T-scores have a mean of 30 ± 10 where higher scores are indicative of better verbal memory. Total T-score differences following study treatment interventions are reported.
Time Frame: At end of each treatment condition (on average 21 days between treatments)
Measure: Mean (Standard Error); unit: T-score
Groups:
- Phenytoin&Hydrocortisone: Examining all participants for the condition in which they took both phenytoin and hydrocortisone.
- Placebo&Placebo: Examining all participants for the condition in which they took placebo for both administrations.
- Phenytoin&Placebo: Examining all participants for the condition in which they took phenytoin and placebo.
- Placebo&Hydrocortisone: Examining all participants for the condition in which they took placebo and hydrocortisone.
Arm/Group | Phenytoin&Hydrocortisone | Placebo&Placebo | Phenytoin&Placebo | Placebo&Hydrocortisone
Number analyzed (Participants) | 15 | 16 | 16 | 15
T-score | 57.76 (0.51) | 56.11 (0.67) | 53.08 (0.45) | 42.76 (2.60)
Statistical Analysis 1: Comparison: Phenytoin&Hydrocortisone vs Placebo&Hydrocortisone; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis
Statistical Analysis 2: Comparison: Phenytoin&Hydrocortisone vs Placebo&Placebo; Test type: Superiority or Other; p = .12, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo&Placebo vs Phenytoin&Placebo; Test type: Superiority or Other; p = .15, Mixed Models Analysis
Statistical Analysis 4: Comparison: Phenytoin&Placebo vs Placebo&Hydrocortisone; Test type: Superiority or Other; p = .10, Mixed Models Analysis

2. Secondary Outcome: Hippocampal Activation Differences Between Treatment Conditions
Time Frame: At the end of each treatment condition
Measure: Mean (Standard Deviation); unit: percentage of BOLD activation
Groups:
- Phenytoin&Hydrocortisone: Participants will take two capsules containing phenytoin tablets (100 mg) by mouth at 0900 hours and 2100 hours (400 mg/day) for a total of three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Beginning two days prior to the imaging (the day after initiating the phenytoin), participants will begin taking 4 tablets containing hydrocortisone (20 mg) also at 0900 hours and 2100 hours (160 mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours.
- PBO&PBO: Participants will take two capsules containing placebo by mouth at 0900 hours and 2100 hours (400 mg/day) for a total of three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Beginning two days prior to the imaging (the day after initiating the placebo), participants will begin taking 4 tablets of placebo also at 0900 hours and 2100 hours (160 mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours.
- Phenytoin&PBO: Participants will take two capsules containing phenytoin tablets (100 mg) by mouth at 0900 hours and 2100 hours (400 mg/day) for a total of three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Beginning two days prior to the imaging (the day after initiating the phenytoin), participants will begin taking 4 tablets containing placebo also at 0900 hours and 2100 hours (160 mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours.
- PBO&Hydrocortisone: Participants will take two capsules containing placebo by mouth at 0900 hours and 2100 hours (400 mg/day) for a total of three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Beginning two days prior to the imaging (the day after initiating the placebo), participants will begin taking 4 tablets containing hydrocortisone (20 mg) also at 0900 hours and 2100 hours (160 mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours.
Arm/Group | Phenytoin&Hydrocortisone | PBO&PBO | Phenytoin&PBO | PBO&Hydrocortisone
Number analyzed (Participants) | 13 | 15 | 15 | 14
percentage of BOLD activation | 1.035 (0.180) | 1.288 (.06) | 1.135 (0.161) | 1.121 (0.144)
Statistical Analysis 1: Comparison: Phenytoin&Hydrocortisone vs PBO&Hydrocortisone; Test type: Superiority or Other; p = .08, Mixed Models Analysis
Statistical Analysis 2: Comparison: Phenytoin&Hydrocortisone vs PBO&PBO; Test type: Superiority or Other; p < .01, Mixed Models Analysis
Statistical Analysis 3: Comparison: PBO&PBO vs Phenytoin&PBO; Test type: Superiority or Other; p < .01, Mixed Models Analysis
Statistical Analysis 4: Comparison: PBO&PBO vs PBO&Hydrocortisone; Test type: Superiority or Other; p = .02, Mixed Models Analysis

3. Secondary Outcome: Para-Hippocampal Activation Differences Between Treatment Conditions
Time Frame: At the end of each treatment condition
Measure: Mean (Standard Deviation); unit: percentage of BOLD activation
Groups:
- PBO&PBO: Participants will take two capsules containing placebo by mouth at 0900 hours and 2100 hours for a total of three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Beginning two days prior to the imaging (the day after initiating the placebo), participants will begin taking 4 tablets containing placebo also at 0900 hours and 2100 hours with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours.
- Phenytoin&PBO: Participants will take two capsules containing phenytoin tablets (100 mg) by mouth at 0900 hours and 2100 hours (400 mg/day) for a total of three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Beginning two days prior to the imaging (the day after initiating the phenytoin), participants will begin taking 4 tablets containing placebo also at 0900 hours and 2100 hours with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours.
- PBO&Hydrocortisone: Participants will take two capsules containing placebo by mouth at 0900 hours and 2100 hours for a total of three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Beginning two days prior to the imaging (the day after initiating the placebo), participants will begin taking 4 tablets containing hydrocortisone (20 mg) also at 0900 hours and 2100 hours (160 mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours.
Arm/Group | Phenytoin&Hydrocortisone | PBO&PBO | Phenytoin&PBO | PBO&Hydrocortisone
Number analyzed (Participants) | 13 | 15 | 15 | 14
percentage of BOLD activation | 1.293 (0.264) | 1.604 (0.315) | 1.464 (0.246) | 1.401 (0.202)
Statistical Analysis 1: Comparison: Phenytoin&Hydrocortisone vs PBO&Hydrocortisone; Test type: Superiority or Other; p = .08, Mixed Models Analysis
Statistical Analysis 2: Comparison: Phenytoin&Hydrocortisone vs PBO&PBO; Test type: Superiority or Other; p < .01, Mixed Models Analysis
Statistical Analysis 3: Comparison: PBO&PBO vs Phenytoin&PBO; Test type: Superiority or Other; p = .11, Mixed Models Analysis
Statistical Analysis 4: Comparison: PBO&PBO vs PBO&Hydrocortisone; Test type: Superiority or Other; p = .06, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Throughout entirety of trial
Groups:
- Phenytoin, Then Hydrocortisone: Placebo, Placebo
  Phenytoin, Dilantin : participants will take two capsules containing phenytoin tablets (100 mg) or identical placebo by mouth at 0900 hours and 2100 hours (400 mg/day) for a total of three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Beginning two days prior to the imaging (the day after initiating the phenytoin or placebo), participants will begin taking 4 tablets containing hydrocortisone (20 mg) or placebo also at 0900 hours and 2100 hours (160 mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours.
- Phenytoin, Then Placebo: Phenytoin, Placebo
  Phenytoin, Dilantin : participants will take two capsules containing phenytoin tablets (100 mg) or identical placebo by mouth at 0900 hours and 2100 hours (400 mg/day) for a total of three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Beginning two days prior to the imaging (the day after initiating the phenytoin or placebo), participants will begin taking 4 tablets containing hydrocortisone (20 mg) or placebo also at 0900 hours and 2100 hours (160 mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours.
- Placebo, Then Hydrocortisone: Hydrocortisone, Placebo
  Phenytoin, Dilantin : participants will take two capsules containing phenytoin tablets (100 mg) or identical placebo by mouth at 0900 hours and 2100 hours (400 mg/day) for a total of three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Beginning two days prior to the imaging (the day after initiating the phenytoin or placebo), participants will begin taking 4 tablets containing hydrocortisone (20 mg) or placebo also at 0900 hours and 2100 hours (160 mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours.
- Placebo, Then Placebo: Hydrocortisone, Phenytoin
  Phenytoin, Dilantin : participants will take two capsules containing phenytoin tablets (100 mg) or identical placebo by mouth at 0900 hours and 2100 hours (400 mg/day) for a total of three days with the last dose at 0900 hours on the day of the imaging (7 doses total). Beginning two days prior to the imaging (the day after initiating the phenytoin or placebo), participants will begin taking 4 tablets containing hydrocortisone (20 mg) or placebo also at 0900 hours and 2100 hours (160 mg/day) with the last dose at 0900 hours on the day of the imaging (5 doses total). The imaging will be performed at 1300 hours.
Arm/Group | Phenytoin, Then Hydrocortisone | Phenytoin, Then Placebo | Placebo, Then Hydrocortisone | Placebo, Then Placebo
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/16 | 1/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/14 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phenytoin, Then Hydrocortisone (N=16) | Phenytoin, Then Placebo (N=16) | Placebo, Then Hydrocortisone (N=14) | Placebo, Then Placebo (N=15)
MRI anxiety (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Physical symptoms manifesting from stress of MRI scan during scan (e.g. difficulty breathing, sweating, tremors, disorientation, etc.)
Pre-existing condition discovered during MRI (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Mega cisterna magna discovered at initial MRI. Determined to be benign.

LIMITATIONS AND CAVEATS:
The sample size in this pilot study was modest; The duration of exposure to hydrocortisone was subacute;

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No